CLINICAL TRIAL: NCT01856283
Title: An Open Label, Single Arm, Phase II Study of Nilotinib 300 mg BID in Newly Diagnosed CP-CML Patients, in Order to Verify Disappearance of CD34+/Lin-Ph+ Cells From Bone Marrow During Treatment
Brief Title: Nilotinib 300 mg BID in Newly Diagnosed CP-CML Patients to Verify Disappearance of CD34+/Lin-Ph+ Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PhilosoPhy34 CAMN107EIT11T
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental): study of nilotinib 300 mg BID
  Interventions: Drug: Nilotinib 300mg BID

INTERVENTIONS:
Drug: Nilotinib 300mg BID — Nilotinib
  Other Names: Nilotinib

SUMMARY:
This is a multicentre, single-arm study of nilotinib 300 mg BID in newly diagnosed patients with CP-CML. This study is designed to establish the disappearance of Ph+ stem cells (CD34+/lin-) in BM during nilotinib treatment.

In addition, in this study the investigators aim to perform Gene Expression Profiling (GEP) of CML enrolled patients using Affymetrix GeneChip Instruments and Software Systems, and Affymetrix GeneChip Human Genome U133 Plus 2.0 (whole human transcriptome analysis) at diagnosis and at 3 different time points during treatment with Nilotinib (after 3, 6, 12 months).

DETAILED DESCRIPTION:
This study is designed to establish the disappearance of Ph+ stem cells (CD34+/lin-) in BM during nilotinib treatment.

The primary efficacy endpoint is to measure the rate of CD34+/lin-Ph+ cells in the BM after 6 months of treatment. In order to obtain this result, BM blood of all enrolled patients will be stored after 6 months of treatment with nilotinib. The isolated CD34+/lin- cells will be employed for standard FISH analysis. These endpoints will be obtained at the central laboratory of Niguarda Ca' Granda Hospital, Milano, Italy.

Secondary endpoints will be reached performing:

* the same analyzes on CD34+/lin- cells at diagnosis, at 3 and 12 months of treatment;
* cytogenetic analysis to estimate the rate of CCyR at 3, 6 and 12 months; this analysis will be performed at each local laboratory;
* molecular analysis to determinate the rate of MR (≤ 10%, ≤ 1%, MMR, MR4,5 IS) at 3, 6 and 12 months in the peripheral blood; the molecular analysis will be performed using the Labnet standardized laboratories in Lombardy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with diagnosis of CP-CML with cytogenetic confirmation of Ph chromosome (9;22) translocation within 3 months of diagnosis
* Patients Ph negative or with variant translocations by standard cytogenetic analysis but Ph positive by FISH, are eligible as well
* Age ≥ 18 years old (no upper age limit given)
* WHO performance status ≤2
* Normal serum levels ≥ LLN (lower limit of normal) of potassium, magnesium, total calcium corrected for serum albumin or phosphorus, or correctable to within normal limits with supplements, prior to the first dose of study medication
* AST and ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to leukaemia
* Alkaline phosphatase ≤ 2.5 x ULN unless considered due to leukaemia
* Total bilirubin ≤ 1.5 x ULN, except know Mb Gilbert
* Serum lipase and amylase ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Written informed consent signed prior to any study procedures being performed

Exclusion Criteria:

* Pre-treatment with HU for > 3 months and with imatinib is not permitted
* Prior accelerated phase including clonal evolution or blast crisis
* Contraindication to excipients in study medication
* impaired cardiac function including any of the following:

  1. LVEF <45%
  2. Complete left bundle branch block
  3. Right bundle branch block plus left anterior hemiblock,bifascicular block
  4. Use of a ventricular-paced pacemaker
  5. Congenital long QT syndrome
  6. Clinically significant ventricular or atrial tachyarrhythmias
  7. Clinically significant resting bradycardia (<50 beats per minute)
  8. QTcF >450 msec on screening ECG.If QTcF >450 msec and electrolytes are not within normal ranges before nilotinib dosing, electrolytes should be corrected and then the patient rescreened for QTcF criterion
  9. Myocardial infarction within 12 months prior to starting nilotinib
  10. Other clinical significant heart disease (e.g. unstable angina,congestive heart failure,uncontrolled hypertension)
* Acute (i.e. within 1 year of starting study medication) or chronic pancreatitis
* Concurrent uncontrolled medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infections,acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol
* Impaired gastrointestinal function or disease that may alter the absorption of study drug (e.g.ulcerative disease,uncontrolled nausea,vomiting and diarrhea,malabsorption syndrome,small bowel resection or gastric by-pass surgery)
* Concomitant medications with potential QT prolongation (see link for complete list: http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm)
* Concomitant medications known to be strong inducers or inhibitors of the CYP450 Isoenzyme CYP3A4:see link for complete list (http://medicine.iupui.edu/flockhart/table.htm)
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding or women of reproductive potential not employing an effective method of birth control.Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of nilotinib.Post menopausal women must be amenorrheic for at least 12 months in order to be considered of non-childbearing potential.Female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Treatment with any haematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF) ≤1 week prior to starting study drug
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
CD34+/lin-Ph+ cells | 6 month
  To measure the rate of CD34+/lin-Ph+ cells in the BM after 6 months of treatment. In order to obtain this result, BM blood of all enrolled patients (see Appendix
  1) will be stored after 6 months of treatment with nilotinib. The isolated CD34+/lin- cells will be employed for standard FISH analysis.

SECONDARY OUTCOMES:
CD34+/lin- cells (composite measure) | 12 month
  Secondary endpoints will be reached performing:
  * the same analyzes on CD34+/lin- cells at diagnosis, at 3 and 12 months of treatment;
  * cytogenetic analysis to estimate the rate of CCyR at 3, 6 and 12 months; this analysis will be performed at each local laboratory; molecular analysis to determinate the rate of MR (≤ 10%, ≤ 1%, MMR, MR4,5 IS) at 3, 6 and 12 months in the peripheral blood; the molecular analysis will be performed using the Labnet standardized laboratories in Lombardy.
  The Outcome Measure indicates that the measure is a composite.

CONTACTS AND LOCATIONS:
Overall Officials: Ester Pungolino, MD, Principal Investigator — Niguarda Ca' Granda Hospital
Locations (17):
- Italy (17):
  - A.O. Ospedale S. Antonio, Gallarate, Milano
  - Ospedale Desio- "Ospedale Civile" di Vimercate, Desio, Carate Brianza, Giussano, Seregno., Vimercate, Milano
  - A.O di Circolo di Busto Arsizio, Busto Arsizio, Varese
  - Ospedali Riuniti Bergamo, Bergamo
  - Spedali Civili Brescia, Brescia
  - Ospedale Valduce, Como
  - Istituti Ospitalieri di Cremona, Cremona
  - A.O Ospedale Lecco, Lecco
  - Ospedale San Raffaele, Milan
  - A.O Sacco, Milan
  - Istituto dei Tumori, Milan
  - Istituto Europeo Oncologia, Milan
  - Ospedale Maggiore Policlinico, Milan
  - Ospedale S. Paolo, Milan
  - S. Gerardo di Monza, Monza
  - Policlinico S.Matteo Pavia, Pavia
  - A.O. Universitaria Fondazione Macchi, Varese